CLINICAL TRIAL: NCT02186275
Title: Randomized Controlled Trial of High Dose Vitamin D in Children With Newly Diagnosed Crohn's Disease for the Prevention of Relapses
Brief Title: The Vitamin D in Pediatric Crohn's Disease
Acronym: ViDiPeC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jantchou Prevost, MD, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JP2014
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Crohn's Disease
Keywords: Crohn; vitamin D; remission; inflammation; tolerance
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 3000 or 4000 UI/day then 2,000 UI/day (Experimental): 3000 UI or 4,000 UI/day as induction therapy (according to weight) for 4 weeks then 2,000 UIday as maintenance therapy for 48 weeks.
  The administration of vitamin D will be considered as an adjunct to conventional therapy (corticosteroids, exclusive enteral nutrition or immunosuppressive agents (ISA)).
  Interventions: Drug: Vitamin D3: 3000 or 4000 UI/day then 2,000 UI/day
- Vitamin D3 800 UI/day then 800 UI/day (Active Comparator): 800 UI/day as induction therapy for 4 weeks, then 800 UI/day as maintenance therapy for 48 weeks. The administration of vitamin D will be considered as an adjunct to conventional therapy (corticosteroids, exclusive enteral nutrition or immunosuppressive agents (ISA)).
  Interventions: Drug: Vitamin D3 800 UI/day then 800 UI/day

INTERVENTIONS:
Drug: Vitamin D3: 3000 or 4000 UI/day then 2,000 UI/day — * Weight at inclusion < 40 kg : 3 capsules of 1000 UI per day at induction and 2 capsules of 1000 UI per day at maintenance.
  * Weight at inclusion ≥ 40 kg : 4 capsules of 1000 UI per day at induction and 2 capsules of 1000 UI per day at maintenance.
  Other Names: Cholecalciferol
  Arms: Vitamin D3 3000 or 4000 UI/day then 2,000 UI/day
Drug: Vitamin D3 800 UI/day then 800 UI/day — * Weight < 40 kg: 2 capsules of 400 UI per day and 1 capsules of placebo at induction and 2 capsules of 400 UI per day at maintenance
  * Weight ≥ 40 kg: 2 capsules of 400 UI per day and 2 capsules of placebo at induction and 2 capsules of 400 UI per day at maintenance
  Other Names: Cholecalciferol
  Arms: Vitamin D3 800 UI/day then 800 UI/day

SUMMARY:
The purpose of this study is to determine if vitamin D as an adjuvant therapy can improve the outcome (i.e. fewer relapses) and the quality of life, including levels of physical activity, in children with newly diagnosed Crohn's disease (CD).

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory condition affecting all segments of the digestive tract from the mouth to the anus. This condition is associated with an increased risk of relapses throughout the course of the disease. Nearly 25% of patients with Crohn's disease are in the pediatric age range. Many epidemiological data are in favor of an increase incidence of pediatric Crohn's disease. Environmental factors could explain this increased incidence. Among them sunlight exposure and vitamin D deficiency have been suggested by many authors.

Recent studies have described how varying doses of oral vitamin D supplementation can alter serum levels of 25 hydroxyvitamin D (25(OH)D), but no study has specifically addressed the question as to whether vitamin D supplementation can alter the rate of relapse/complications and/or quality of life in children diagnosed with CD.

Current treatments of CD at diagnosis are effective around the time of diagnosis, but in the short and long term, some of these therapies are inefficient or lead to allergic or intolerance reactions. Altogether the rate of relapses in the year after diagnosis is significant. Thus, different therapeutic approaches must be investigated with the aim of lowering the burden of the disease.

From November 2012 to July 2013, we conducted an open label pilot cohort study aiming to investigate the bioavailability and tolerance of high doses of vitamin D3 (3,000 IU or 4,000 IU per day) administered orally as an adjunct therapy in 20 children with newly diagnosed pediatric CD (http://clinicaltrials.gov/ct2/show/NCT01692808). Data from laboratory studies, observational research and pilot trials taken together suggest that vitamin D can be of great importance in the genesis and progression of CD. Vitamin D deficiency could be a true risk factor for disease occurrence and/or relapses. The results of our pilot study demonstrate that in children with active CD at diagnosis, a daily dose of 4,000 IU of vitamin D is well tolerated and quickly increases the blood levels of 25OHD3 to 100 nmol/L or above in 100% of children with CD at diagnosis. Moreover a maintenance dosage of 2,000 IU a day is required (and sufficient) for maintaining this target over several months. Currently there is no adequately powered study in the pediatric CD population exploring the relationship between vitamin D therapy at diagnosis and CD outcomes.

We propose a randomized controlled trial (RCT) to study the efficacy of high-dose oral vitamin D, as adjunct therapy, in children with newly diagnosed CD, to reduce the relapse rate and to improve patients' quality of life.

Primary Efficacy End Point: The proportion of patient with at least one relapse 52 weeks after randomization.

Secondary efficacy endpoint: Quality of life scores, Cumulative steroid dose, Time to first relapse, Duration of corticotherapy, Number of relapses, Number of hospitalizations Safety Endpoint : incidence of hypercalcemia (defined as a corrected serum calcium level >2.65 mmol/L), incidence of hypercalciuria (defined as urinary calcium to creatinine molar ratio ≥1.50), incidence of supra-optimal levels of 25OHD3 as defined by a serum level ≥ 250 nmol/L, rate of study discontinuation due to hypercalcemia or hypercalciuria.

Efficacy Variable: Occurrence of relapse, Time to relapse, Change in QoL score from baseline to 26 weeks, 52 weeks. Change in physical activity score from baseline to 26 weeks, 52 weeks.

ELIGIBILITY:
Eligibility Criteria:

- Diagnosis of CD by the usual clinical, endoscopic and histological criteria and classified according to the Paris classification

Inclusion Criteria:

* Age at randomization between 9 and 18 years inclusively
* Interval between diagnosis and randomization between 2 weeks and 6 months after the diagnosis
* Pediatric Crohn's Disease Activity Index (PCDAI) ≤ 30 at inclusion
* Concurrent treatment with corticosteroids and/or enteral nutrition and/or thiopurines (azathioprine, 6-mercaptopurine) and/or methotrexate and/or 5-aminosalicylic acid (5-ASA) and/or TNF-α inhibitors (Infliximab, Adalimumab).

Exclusion Criteria:

* Patient diagnosed with severe complex perianal fistulizing CD (defined as the presence at diagnosis of a high intersphincteric, transsphincteric, extrasphincteric, or suprasphincteric complex perianal fistula)
* Known chronic liver cholestasis (defined by an elevation of conjugated bilirubin and/or gamma glutamyl transferase > 3 upper limit normal)
* Known renal dysfunction requiring chronic dialysis or creatinine ≥ 100 micromol/L.
* Known congenital bone disease
* Known cystic fibrosis or other exocrine pancreatic insufficiency.
* Currently treated with anticonvulsants metabolized through cytochrome P-450
* Unable to take oral capsule form.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one relapse within 52 weeks after randomization in the trial. | within 52 weeks after inclusion in the study
  A relapse is defined as the occurrence of clinical symptoms (> 2 bowel movements per day, abdominal pain, fever, weight loss, perianal disease or extra-intestinal symptoms) and a pediatric Crohn's disease Activity Index (PCDAI) > 30.
  The PCDAI is a validated and reproducible tool that was developed by consensus at a meeting of pediatric (Inflammatory bowel disease) IBD experts and subsequently validated in 12 North American institutions. It includes 11 domains, with clinical symptoms, physical examination, laboratory parameters, and growth.
  The PCDAI score can range from 0-100, with higher scores signifying more active disease. A score < 10 is consistent with inactive disease; 11-30 indicates mild disease; > 30 suggests moderate to severe disease. The PCDAI has been used in many pediatric trials.

SECONDARY OUTCOMES:
the lapse of time from randomization to first relapse | from randomization to first relapse
the number of relapses per patient per year | within 52 weeks after randomization in the trial
the duration of corticotherapy | between randomization and 52 weeks later
The number of CD related hospitalizations | between randomization and 52 weeks later
The quality of life | at 26 weeks and 52 weeks
  as measured by the IMPACT III questionnaire. IMPACT III is a validated questionnaire that assesses disease-related quality-of-life in multiple domains of care in pediatric IBD (bowel symptoms; systemic symptoms; emotional functioning; functional/social impairment; body image; test-treatments). Overall scores for IMPACT III range from 35 to 175 with higher scores associated with better quality of life

OTHER OUTCOMES:
Change in the level of physical activities | between randomization and 52 weeks later
  As measured by the Canadian Health Measures Survey (CHMS) - Children's Physical ActivityQuestionnaire
Changes in bone mineral density | between randomization and 52 weeks later
  As assessed by dual energy X-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Prevost Jantchou, MD, Principal Investigator — St. Justine's Hospital
Locations (10):
- Canada (10):
  - Edmonton Clinic Health Academy, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Health Science Center Pediatric, Winnipeg, Manitoba
  - Janeway Children's Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Hospital for Sick Childrens, Toronto, Ontario
  - Montreal Children's Hospital (Montreal)., Montreal, Quebec
  - Ste-Justine hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire Laval, Québec